CLINICAL TRIAL: NCT04874519
Title: Fibrolamellar Carcinoma Global Dynamic Registry
Brief Title: Registry to Collect Health Information Related to Fibrolamellar Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-543
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Fibrolamellar Cancer; FLC; Liver Cancer
Keywords: fibrolamellar cancer; liver cancer; 20-543; Memorial Sloan Kettering Cancer
MeSH Terms: conditions — Fibrolamellar hepatocellular carcinoma; Liver Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Fibrolamellar Carcinoma/FLC: Participants will have a personal history of histologically proven fibrolamellar carcinoma (clinical or radiographical suspicion of FLC must be confirmed at MSK or an external hospital)
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — The questionnaire will be completed at the time of enrollment, every month, and at the end of study. Regardless of current interventions or lack of, assessments will be completed at enrollment and then monthly for a total of 18 months. In order to provide reasonable flexibility to participants, physicians, and study teams, the assessments can be completed within 30 days of the last assessment. The next month will be recalculated based on last reporting date.

SUMMARY:
The purpose of this study is to collect information about people with fibrolamellar cancer (FLC). This study is a registry of people with FLC around the world. This study will involve collecting information about participants, their medical history and the regular medical care they receive for FLC. The study will not provide treatment for your cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 years or older.
* Personal history of histologically proven fibrolamellar carcinoma (clinical or radiographical suspicion of FLC must be confirmed at MSK or an external hospital)
* Participants must have access to electronic devices that meet the following minimum requirements:

  * Ability to connect to the internet
  * Capability of running modern internet browers (such as Google Chrome, Internet Explorer, Safari, or Mozilla Firefox).
* Participants must have a google account

Exclusion Criteria:

* Participants residing in the European Union (EU).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential research subjects may also be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan Kettering Cancer Center (MSKCC). If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. Potential subjects contacted by their treating physician will be referred to the investigator/research staff of the study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Build a Fibrolamellar Cancer/FLC registry | 18 months
  To build a registry of Fibrolamellar Cancer/FLC through patient reported information, that could be studied further in future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan Abou-Alfa, MD, MBA, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org